CLINICAL TRIAL: NCT02158793
Title: Craniomaxillofacial Allotransplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was determined that the study would be integrated into the standard clinical care.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00550
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Facial Injuries
Keywords: face transplant; Craniomaxillofacial Allotransplantation; facial disfigurement; facial trauma
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Face Transplant recipient (Experimental): Single Arm study, all participants will receive Craniomaxillofacial allotransplantation
  Interventions: Procedure: Craniomaxillofacial allotransplantation

INTERVENTIONS:
Procedure: Craniomaxillofacial allotransplantation — Transplantation of donor face

SUMMARY:
The purpose of this study is to perform face transplants on people who have suffered severe facial trauma with tissue and functional loss; and evaluate the acceptance and function of the transplanted tissue. The aim of the transplant is to provide patient a more normal appearance . Additionally we aim to restore functioning, movement, and sensation of their face including that of the lips, mouth, and eyes.

DETAILED DESCRIPTION:
This study is to perform facial transplants in patients with severe facial deformities or facial wounds from traumatic injuries. The transplant is to help reconstruct a person's damaged face. The aim of the transplant is to provide patient a more normal appearance . Additionally we aim to restore functioning, movement, and sensation of their face including that of the lips, mouth, and eyes.

There are some procedures in plastic and reconstructive surgery that can repair the look of a patient's face, but often can't replace the movement and use of the face. Currently, patients with severe facial deformities would undergo several reconstructive surgeries with their own tissues, called autologous transplant. Conventional reconstruction method requires multiple surgeries in order to form and shape the transplanted tissue. Because this type of reconstruction is limited, it does not provide a reliable return in function, sensation, and appearance for the damaged parts of the face.

This study uses a composite tissue allograft , or face transplant from a donor who is brain dead such as in heart, kidney and liver transplants. The damaged parts of the face could return movement as well. Transplanted patients are required to take lifelong immunosuppression drugs which have risks, which are still a consideration when deciding to choose this option for correcting severe facial deformities.

We will conduct the surgery and prospectively follow the patient to monitor signs of rejection of the transplanted face. Additionally, patients will be constantly evaluated for clinical and functional outcomes and ensure that optimal results are achieved.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated all required IRB approved consent forms
* Male or female recipient between the ages of 18-64 years. * Recipients do not need to be same gender as donor*
* Facial composite tissue defect requiring facial transplantation as determined by the treating Plastic and Reconstructive Surgeon. Inclusive facial functional subunit tissue loss. Including but not limited to irreparable peri-oral, peri-orbital, and peri-nasal damage.
* Patient has been encouraged to seek a second opinion from a Plastic Surgeon with specialized focus in facial reconstruction.
* Willingness to participate in ongoing psychiatric, psychological and social work evaluations prior to and post-transplant surgery
* The subject is able to complete pre-transplant examination and screening procedures.
* Patient has been approved by Patient Selection Committee for placement on the recipient waiting list
* The subject is willing to continue immunosuppression regimen as directed by treating physician.
* Subject is willing and able to return to follow-up visits as described in treatment plan.
* Subjects must have autogenous tissue options available for reconstruction in event of graft failure.
* Normal GFR (glomerular filtration rate) >60
* Negative pregnancy test within 48hrs of transplant for women of childbearing age and who agree to use a reliable form of contraception for one year following transplant.

Exclusion criteria:

* Subject has an uncontrolled infection
* Serious co-morbidities
* Positive serology for HIV; Hepatitis B/C Antigen
* Active malignancy within 5 years with the exclusion of non-melanoma
* Subject has active substance abuse/ alcoholism
* Active Severe Psychiatric Illness
* Cognitive limitations affecting the patient's ability to provide informed consent
* Recent history of medical nonadherence
* Unstable social situation as evidence by lack of stable housing and/or lack of a supportive significant other.
* Recent history of medical non-adherence.
* Lack of stable housing and/or supportive significant other/caregiver throughout all phases of the study
* Currently active smoker within 1 year
* Subjects with any cognitive deficits related to a TBI (traumatic brain injury) and or any organic neurological disorders will not be considered for this protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the success of the face transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  We will measure the restoration of function, sensation, and appearance of the transplanted facial segment.
  These will be measured using various multi-disciplinary evaluations including swallow studies, photography, speech therapy evaluation, Occupational therapy evaluation, electromyogram (EMG) , Nerve Conduction Study (NCS), CT Angiogram, Functional ( Magnetic Resononance Image) MRI, vision exams, pathology samples to check for rejection, Blood tests

SECONDARY OUTCOMES:
Evaluate psychological effects of receiving a face transplant | Monthly for 6 months, every 6 months for 2 years, then annually until year 5
  Psychological outcome will be measured using patient reported outcome tools such as MoCA; BIDQ; SF-36; PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rodriguez, MD, DDS, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States